CLINICAL TRIAL: NCT00487734
Title: Effect of Testosterone Replacement on Insulin Resistance in Hypogonadal, Non-obese Men With Metabolic Syndrome
Brief Title: Effect of Testosterone Replacement on Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGuire Research Institute (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01274
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Metabolic Syndrome; Hypogonadism
Keywords: Metabolic Syndrome; Hypogonadism; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Hypogonadism; Insulin Resistance | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects in this arm will receive testosterone gel
  Interventions: Radiation: Testosterone gel
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo for testosterone gel

INTERVENTIONS:
Radiation: Testosterone gel — testosterone gel, applied daily. Dosed to achieve testosterone level <500 ng/dL. Possible doses include 2.5g, 5g, 7.5g or 10g gel packets.
  Other Names: Androgel
  Arms: 1
Drug: Placebo for testosterone gel — Placebo gel, 2.5g for each gel packet
  Arms: 2

SUMMARY:
This study aims to determine whether testosterone replacement improves insulin sensitivity in non-obese men with low testosterone and the metabolic syndrome. The metabolic syndrome includes three of the following five conditions, 1) an elevated blood pressure (greater than 130/85), 2) a triglyceride level greater than 150 mg/dl, 3) an HDL-cholesterol less than 40 mg/dl, 4) glucose levels greater than 100 mg/dl, and 5) a waist measurement greater than 40 inches.

DETAILED DESCRIPTION:
In this proposal, we will examine the relationship between hypogonadism and insulin sensitivity. The strongest relationship between hypogonadism and insulin resistance appears to reside in men with the metabolic syndrome who have a normal BMI. The causal relationship between these two conditions is unknown. Therefore, we propose to determine if testosterone replacement in hypogonadal non-obese men with metabolic syndrome will improve insulin sensitivity. Data obtained from this preliminary investigation, will hopefully result in a hypothesis that can be tested in a larger, more rigorous trial in the future.

ELIGIBILITY:
Inclusion Criteria: (subjects must meet both criteria)

* Metabolic syndrome (have 3 out of the following 4 criteria):

  1. BP > 130/85 or on antihypertensive therapy
  2. Fasting glucose > 100 mg/dl
  3. Fasting TG > 150 mg/dl or on a triglyceride lowering agent (fenofibrate, gemfibrozil, niacin in doses of >= 500 mg/day, or fish oils in doses of >=2000mg DHA+EPA)
  4. Fasting HDL-C < 40 mg/dl Note that the waist circumference will not be used as one of the criteria for the metabolic syndrome for this study because we are studying non-obese subjects.
* Total Testosterone less than 300 ng/dl

Exclusion Criteria:

* Women.
* Men less than 20 years of age.
* BMI > or = to 30 kg/M2.
* Use of testosterone preparations within 1 year of the screening visit
* Use of hypoglycemic medications within the previous 3 months.
* Fasting blood glucose > 126 mg/dl.
* The following men will be excluded because of the potential safety issues in the placebo treated group:

  1. Creatinine greater than 1.4 mg/dl
  2. Triglyceride levels greater than 500 mg/dl
  3. HDL-C levels less than 20 mg/dl
  4. Blood pressure greater than 160/90
* The following men will be excluded because of the potential side effects of testosterone therapy:

  1. Men greater than 65 years of age
  2. International prostate symptom score >19
  3. PSA greater than 2.5
  4. History of benign prostatic hypertrophy
  5. History of prostate cancer
  6. Abnormal digital rectal exam
  7. Hg greater than 16 mg/dl or Hct greater than 48%
  8. peripheral edema

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity as measured by HOMA-IR | 18 weeks

SECONDARY OUTCOMES:
Changes in parameters of the Metabolic Syndrome | 18 weeks
Changes in body composition | 18 weeks
Changes in total and high MW adiponectin levels | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sonja K Fredrickson, MD, Principal Investigator — Hunter Holmes McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States